CLINICAL TRIAL: NCT03202706
Title: Use of Biopsies of Abdominal Subcutaneous Fat to Study the Role of the Activation of Endocannabinoid 1 Receptors (CB1R) on Adipocyte Glucolipid Metabolism
Acronym: CB1R
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: VERGES 2015
Record Dates: First submitted 2017-06-21; First posted 2017-06-28 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Hernia Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients
  Interventions: Procedure: Samples of adipose tissue

INTERVENTIONS:
Procedure: Samples of adipose tissue — Samples of visceral and subcutaneous adipose tissue collected during hernia surgery

SUMMARY:
Obesity is associated with hyperactivation of the endocannabinoid system, and its inhibition by the administration of CB1 receptor (CB1R) antagonists, leads to a decrease in food intake, weight loss and an improvement in metabolic parameters. Even though the reduction in food intake following central CB1R inactivation seems to be the principal cause of weight loss and the improvement in metabolic parameters, several studies in animals and humans have indicated that peripheral CB1R could also be implicated in the regulation of glucolipid metabolism. As a result, it has been suggested that the long-term beneficial effects of inactivation of the endocannabinoid system are due to both central effects on food intake and peripheral effects involving adipose tissue, the liver, skeletal muscle and the pancreas. It appears essential to determine the role of CB1R located in peripheral tissues and in particular in adipose tissue, which plays an active role in maintaining glucolipid homeostasis. The experiments conducted in this project consist in studying in biopsies of abdominal subcutaneous fat whether activation of adipocyte CB1R modifies adipocyte metabolism by determining the mechanisms. The investigators hypothesize that activation of CB1R in adipose tissue will lead to the stimulation of lipolysis dependent on the alteration of the insulin signal, and therefore that inactivation of the endocannabinoid system by blocking peripheral CB1R could constitute a therapeutic approach to improve obesity-related insulin resistance and dyslipidaemia.

ELIGIBILITY:
healthy subjects

Inclusion Criteria:

* men aged 18 to 70 years
* persons who have provided oral consent
* persons undergoing surgery for hernia

Exclusion Criteria:

* persons without health insurance cover
* BMI > 30
* diabetes
* associated diseases: cancer, chronic inflammatory diseases
* adults under guardianship

obese subjects

Inclusion Criteria:

* men aged 18 to 70 years
* BMI > 30
* persons who have provided oral consent
* persons undergoing surgery for hernia

Exclusion Criteria:

* persons without health insurance cover
* diabetes
* associated diseases: cancer, chronic inflammatory diseases
* adults under guardianship

diabetic obese subjects

Inclusion Criteria:

* men aged 18 to 70 years
* type 2 diabetic not treated with Insulin or GLP-1 agonist
* BMI > 30
* persons who have provided oral consent
* persons undergoing surgery for hernia

Exclusion Criteria:

* persons without health insurance cover
* associated diseases: cancer, chronic inflammatory diseases
* adults under guardianship

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing surgery for hernia
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2016-02-24 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-01-07 (Actual)

PRIMARY OUTCOMES:
Glucolipid metabolism analysis in human abdominal subcutaneous and visceral fat | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France